CLINICAL TRIAL: NCT03767894
Title: MyHand: An Active Hand Orthosis for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Wallace H. Coulter Foundation (Other); U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joel Stein, MD, Simon Baruch Professor of Physical Medicine and Rehabilitation, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAP8752; IIS-1526960 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2018-11-14; First posted 2018-12-07 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: Hand orthosis; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Masking Description: Subjects are assessed by an independent therapist. The therapist is not blinded to the control mechanism used during treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MyHand orthosis (Experimental): Subjects are trained to control and use the MyHand orthosis either with a shoulder harness or an electromyography (EMG) band. The MyHand orthosis aims to aid in fine motor skills such as picking up and holding items of varying shape, size and weight.
  Interventions: Device: EMG Band; Device: Shoulder harness

INTERVENTIONS:
Device: EMG Band — The MyHand orthosis provides tension to the digits to open the fingers on demand. This group will wear an EMG band to control and activate the MyHand orthosis.
Device: Shoulder harness — The MyHand orthosis provides tension to the digits to open the fingers on demand. This group will wear a shoulder strap to control and activate the MyHand orthosis, either with shoulder elevation or shoulder depression.

SUMMARY:
This study seeks to explore the efficacy of several control mechanisms for the device and the impact of a device training program on its utility as a neuroprosthetic and training tool for upper limb recovery.

DETAILED DESCRIPTION:
Hand rehabilitation through occupational therapy is critical for many stroke survivors, but it is also greatly limited by insurance coverage, shortage of therapists, and logistic constraints. To address this, stroke patients need a rehabilitation method they can use on their own, without direct clinical supervision, and for activities of daily living. MyHand is a wearable and active hand orthosis consisting of a glove and forearm splint, equipped with actuators and tendons which connect to the fingers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age
* History of stroke resulting in significant upper limb impairment
* Full passive range of motion
* Gross control of the proximal upper extremity
* Lacks timely grasp/release
* No more than moderate flexor tone
* Intact cognition

Exclusion criteria include:

* Other Neurological/orthopedic disorders
* Excessive spasticity/contracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MyHand Orthosis: Subjects are trained to control and use the MyHand orthosis either with a shoulder harness or an EMG band. The MyHand orthosis aims to aid in fine motor skills such as picking up and holding items of varying shape, size and weight.
  EMG Band: The MyHand orthosis provides tension to the digits to open the fingers on demand. This group will wear an EMG band to control and activate the MyHand orthosis.
  Shoulder harness: The MyHand orthosis provides tension to the digits to open the fingers on demand. This group will wear a shoulder strap to control and activate the MyHand orthosis, either with shoulder elevation or shoulder depression.
Period: Overall Study
Arm/Group | MyHand Orthosis
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 11 participants participated in and completed the intervention protocol.
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 52 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Type of Stroke [Count of Participants; unit: Participants]
  Ischemic Stroke | 9
  Hemorragic Stroke | 1
  Unknown Type (by participant) | 1

OUTCOME MEASURES:

1. Primary Outcome: Score on Action Research Arm Test (ARAT)
Description: The ARAT is a 19-item measure that assesses upper limb functioning. The ARAT is divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from 0 (cannot perform) to 3 (normal performance). Scores on the ARAT range from 0-57 points, with higher scores indicating better performance.
Time Frame: Baseline; Post-test at Week 4
Population: Only the 11 subjects that completed the study were included in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
score on a scale
  Baseline | 13.46 (2.184)
  Post Unassisted (week 4) | 14.82 (2.148)
  Post Assisted (week 4) | 13.09 (1.43)
Statistical Analysis 1: Comparison: MyHand Orthosis; Baseline scores compared to Post Unassisted condition (ARAT performed unassisted/without the use of the MyHand device); Test type: Other — Descriptive analysis (paired sample t-test); p = 0.24, t-test, 2 sided — a priori threshold: p<0.05 p-value is adjusted for multiple comparisons using Bonferroni correction; Adjustment for p-value is 2; Mean Difference (Final Values) = 1.36
Statistical Analysis 2: Comparison: MyHand Orthosis; Post Unassisted condition (ARAT performed unassisted/without the use of the MyHand device) compared to Post Assisted condition (ARAT performed assisted with the use of the MyHand device); Test type: Other — Descriptive analysis (paired sample t-test); p = 0.207, t-test, 2 sided — a priori threshold: p<0.05 p-value is adjusted for multiple comparisons using Bonferroni correction; Adjustment for p-value is 2; Mean Difference (Final Values) = -1.72

2. Primary Outcome: Score on the Upper Extremity Component of the Fugl-Meyer Scale (UEFM)
Description: The Fugl-Meyer (FM) Assessment of Motor Recovery evaluates and measures recovery in post-stroke hemiplegic patients. The FM uses a 3-point ordinal scale from 0 (cannot perform) to 2 (performs fully). The FM has 5 domains with a maximum score of 226 points. Subscales can be administered with out using the full FM. The Upper Extremity component (UEFM) consists of 33 items with a score range of 0-66. Higher score indicate better performance.
  Please note: An a prior decision was made to only perform the UEFM once at post-testing: post test without robotic assistance. The UEFM assesses capacity of the arm primarily through gross motor tasks, and comparatively few grasping and pinching tasks. Thus, it was presumed that robotic assistance would have minimal influence on UEFM scores. In other words, the UEFM was intended as a outcome measure to primarily evaluate the rehabilitative effects of training with the device, as opposed to evaluating the assistive capacity of using the device.
Time Frame: Baseline; Post-test at Week 4
Population: Only the 11 subjects that completed the study were included in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
score on a scale
  Baseline | 25.36 (1.521)
  Post Unassisted (week 4) | 28 (1.854)
Statistical Analysis 1: Comparison: MyHand Orthosis; Baseline scores compared to Post Unassisted condition (UEMF performed unassisted/without the use of the MyHand device); Test type: Other — Descriptive analysis (paired sample t-test); p = 0.026, Paired sample T-test — a priori threshold: p<0.05; 2-tailed; Mean Difference (Final Values) = 2.64

3. Secondary Outcome: Score on Modified Ashworth Scale (MAS)
Description: The Ashworth or Modified Ashworth Scale (MAS) is a measure of spasticity originally developed as a simple clinical classification to assess the anti-spastic effects of carisoprodol in multiple sclerosis. It is rated on a 5-point nominal scale using subjective clinical assessments of tone ranging from 0 (no increases in tone) to 4 (limb rigid in flexion/extension or abduction/adduction).
  Please note: MAS is officially scored on a 5-point scale that includes "1+" (full range: 0, 1, 1+, 2, 3, 4). However non-numeric scores are not allowable in the Outcome Measure Data Table. Therefore, the scores were transformed from a 0-4 scale (including 1+) to a 0-5 scale (excluding 1+). The reported medians for all but Finger Flexors were not impacted by the scale transformation. Finger Flexor median is reported as 2 in the Outcome Measure Data Table, but this can be understood as a true median of 1+ if using the original MAS scoring scale.
Time Frame: Baseline
Population: Baseline scores on MAS. Only the 11 subjects that completed the study were included in this analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
score on a scale
  Elbow Flexors (baseline) | 1 [0 to 5]
  Elbow Extensors (baseline) | 1 [0 to 5]
  Wrist Flexors (baseline) | 1 [0 to 5]
  Wrist Extensors (baseline) | 0 [0 to 5]
  Finger Flexors (baseline) | 2 [0 to 5]
  Finger Extensors (baseline) | 0 [0 to 5]

4. Secondary Outcome: Score on Box and Blocks Test (BBT)
Description: The BBT measures unilateral gross manual dexterity using blocks and a 2-compartment box. At the start, there are 150 blocks in one compartment and the score represents the number of blocks transferred from one compartment to the other compartment in 60 seconds. Each hand is scored separately, however only scores for the impaired (hemiplegic) hand are reported. Scores can range from 0-150, with higher scores indicating better performance of manual dexterity.
Time Frame: Baseline; Post-test at Week 4
Population: Only the 11 subjects that completed the study were included in this analysis.
Measure: Mean (Standard Error); unit: Blocks
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
Blocks
  Baseline | 47 (2.289)
  Post Unassisted (week 4) | 35 (1.843)
  Post Assisted (week 4) | 24 (0.585)
Statistical Analysis 1: Comparison: MyHand Orthosis; Baseline scores compared to Post Unassisted condition (BBT performed unassisted/without the use of the MyHand device) of the impaired (hemiparetic) hand; Test type: Other — Descriptive analysis (paired Wilcoxon); p = 0.442, Wilcoxon (Mann-Whitney) — a priori threshold: p<0.05 p-value is adjusted for multiple comparisons using Bonferroni correction; Adjustment for p-value is 2; Mean Difference (Final Values) = -1.09
Statistical Analysis 2: Comparison: MyHand Orthosis; Post Unassisted condition (BBT performed unassisted/without the use of the MyHand device) compared to Post Assisted condition (BBT performed assisted with the use of the MyHand device); Test type: Other — Descriptive analysis (paired Wilcoxon); p = 1.0, Wilcoxon (Mann-Whitney) — a priori threshold: p<0.05 p-value is adjusted for multiple comparisons using Bonferroni correction; Adjustment for p-value is 2; Mean Difference (Final Values) = -1

5. Secondary Outcome: Number of Participants Completing Treatment Protocol
Description: The number of participants who completed the full treatment protocol (12 training sessions).
Time Frame: 4 Weeks
Population: Number of participants who completed the treatment protocol (12 sessions). Only the 11 subjects that completed the study were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
Participants | 11

6. Secondary Outcome: Total Number of Adverse Events During Intervention
Description: All adverse events will be tracked during the course of the intervention. The Principal Investigator will review any event and assess it as either adverse or non-significant.
Time Frame: 4 Weeks
Population: Number of participants who experienced adverse events. Only the 11 subjects that completed the study were included in this analysis.
Measure: Number; unit: adverse events
Arm/Group | MyHand Orthosis
Number analyzed (Participants) | 11
adverse events | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | MyHand Orthosis
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03767894/Prot_SAP_000.pdf